CLINICAL TRIAL: NCT03476382
Title: The Use of Bone Growth Stimulators for Osteoarthritis of the Knee.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coastal Carolinas Integrated Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCIM 0001
Record Dates: First submitted 2018-03-18; First posted 2018-03-26 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Osteo Arthritis Knee
Keywords: Osteoarthritis; Knee; Bone Growth Stimulators; Rheumatic Diseases; Musculoskeletal Diseases; Joint Diseases; Arthritis
MeSH Terms: conditions — Osteoarthritis; Rheumatic Diseases; Musculoskeletal Diseases; Joint Diseases; Arthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Experimental Group (Experimental): Participants use active Ultrasound Bone Growth Stimulator device according to Investigational Protocol.
  Interventions: Device: Ultrasound Bone Growth Stimulator

INTERVENTIONS:
Device: Ultrasound Bone Growth Stimulator — Active device emits ultrasound signals.

SUMMARY:
The hypothesis of this study is that since osteoarthritis of the knee is primarily a bone disease where the joint changes are secondary, and bone growth stimulators function to decrease intraosseous venous congestion and remodel bone, then there is a potential benefit for the treatment of osteoarthritis of the knee with bone growth stimulators.

DETAILED DESCRIPTION:
The hypothesis of this study is based on the knowledge that osteoarthritis of the knee is primarily a bone disease, and the joint changes are secondary. Bone growth stimulators function to alleviate intraosseous venous congestion through the process of bone remodeling. The working hypothesis is that alleviation of intraosseous venous congestion leads to improved delivery of nutrition to the tissue to support the health of the bone with improvement in biomechanics leading to clinical improvement. Venous congestion is measured with intraosseous pressure. Additional objective evidence of biomarkers of bone metabolism as well as measurements of subjective questionnaires can provide evidence of benefit.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have diagnosis of osteoarthritis of the knee with radiographic evidence of joint space narrowing, Kellgren-Lawrence Classification grade Grade 3 or 4.
2. Subjects must discontinue corticosteroids administered by any route except intranasal spray, steroid- containing ophthalmic solutions and anti-asthmatics.
3. Subjects must speak English.
4. Subject must be willing and able to sign an informed consent document.
5. Subjects must be willing and able to comply with all study procedures for the duration of the clinical study.

Exclusion Criteria:

1. Subjects with a diagnosis of inflammatory arthritis such as rheumatoid arthritis, gout, joint infection, Lyme disease, or systemic lupus erythematosus.
2. Subjects with a diagnosis of secondary arthritis such as acromegaly, Charcot's arthropathy, hemochromatosis, or Wilson's disease.
3. Subjects who have had an injury to the index knee within 6 months of starting treatment.
4. Subjects must NOT have had arthroscopy within 8 weeks of starting treatment.
5. Subjects must NOT have had viscosupplementation within 8 weeks of starting treatment.
6. Subjects who plan to have surgery on the target knee within the study period.
7. Subjects with surgical metallic hardware in the target knee.
8. Subjects who are unwilling or unable to adhere to the follow up schedule and procedures.
9. Subjects who are pregnant.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2018-11-15 (Actual); Study Completion 2018-11-15 (Actual)

PRIMARY OUTCOMES:
Intraosseous Venous Congestion measured by Intraossous Pressure. | 14 weeks
  Statistically significant decrease in intraosseous pressure following treatment.

SECONDARY OUTCOMES:
Human Matrix Metalloproteinase-3 (MMP-3) | 14 weeks
  Statistically significant decrease in the biomarker MMP-3
C- telopeptide. | 14 weeks
  Statistically significant decrease in the biomarker C- telopeptide.
Change over time in WOMAC score. | 14 weeks
  The primary outcome variables are a statistically significant improvement in Western Ontario and McMaster Universities Arthritis Index (WOMAC) scores.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Willeford, MD, Study Chair — Coastal Carolinas Integrated Medicine; Sierra Willeford, Principal Investigator — Coastal Carolinas Integrated Medicine; Breanna Willeford, Principal Investigator — Coastal Carolinas Integrated Medicine
Locations (1):
- Coastal Carolinas Integrated Medicine, Supply, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No